CLINICAL TRIAL: NCT00872521
Title: A Phase II Trial of Bortezomib, Doxorubicin and Dexamethasone (PAD) Induction Therapy in Patients With Untreated Multiple Myeloma (MM), Stratified for Markers of Bortezomib Resistance
Brief Title: A Study of Efficacy of Treatment With Bortezomib (in Combination With Doxorubicin and Dexamethasone) in Previously Untreated Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen-Cilag Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015640; 26866138MMY2059 (Other: Janssen-Cilag Pty Ltd, Australia); PIMMS Trial (Other: Janssen-Cilag Pty Ltd, Australia)
Record Dates: First submitted 2009-03-27; First posted 2009-03-31 (Estimated); Results first posted 2013-05-07 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; transplant eligible; doxorubicin; dexamethasone; bortezomib; bortezomib resistance; PAD induction; PIMMS Trial
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bortezomib; doxorubicin; dexamethasone (Experimental): PAD induction Open Label Treatment: Four 21-day Treatment Cycles Bortezomib 1.3 mg/m2 i.v. (D1 4 8 & 11) Doxorubicin 20 mg/m2 i.v. (D1 & 4) Dexamethasone 20 mg p.o. (D1 2 4 5 8 9 11 & 12)
  Interventions: Drug: PAD induction

INTERVENTIONS:
Drug: PAD induction — Open Label Treatment:
  Four 21-day Treatment Cycles Bortezomib 1.3 mg/m2 i.v. (D1, 4, 8 & 11), Doxorubicin 20 mg/m2 i.v. (D1 & 4), Dexamethasone 20 mg p.o. (D1, 2, 4, 5, 8 , 9, 11 & 12)

SUMMARY:
The purpose of this study is to determine efficacy of treatment with bortezomib (in combination with doxorubicin and dexamethasone) in previously untreated patients with Multiple Myeloma.

DETAILED DESCRIPTION:
This is an open-label, single-arm, multicentre study which will enroll approximately 105 patients. Open-label means all people involved in the study know the identity of the intervention. Single-arm means there is one group of patients, all receiving the same treatment. Four 21-day cycles of a combination of bortezomib i.v. (intravenous) 1.3 mg/m2 (Days 1, 4, 8 and 11), doxorubicin i.v. 20 mg/m2 (days 1 and 4) and dexamethasone p.o. (by mouth) (days 1, 2, 4, 5, 8, 9, 11 and 12) (PAD) will be given. Patients will be discontinued if disease progresses, or unacceptable treatment-related toxicity occurs. Following PAD treatment, patients will have peripheral blood stem cells (PBSC) collected, and an autologous stem cell transplant (ASCT) will be performed. Patients will then make monthly visits to the Study Doctor until 1 year after start of treatment, and attend a final follow-up visit at 2 years. Efficacy assessment of response to PAD will be made using the International Myeloma Working Group (IMWG) criteria. The primary outcome is to compare the overall response rate following 4 cycles of PAD induction therapy between patients with and without extra copies of the long arm of the first chromosome (1q21) measured by fluorescent in situ hybridisation (FISH) in their marrow at baseline. Patient reported outcomes will be assessed using the AQoL (Assessment of Quality of Life). Safety will be evaluated throughout the study by assessment of adverse events including changes in physical examination, concomitant medication, ECOG (Eastern Cooperative Oncology Group) scores, vital signs and clinical laboratory findings. A sample size of 105 provides 80% power (a=0.05) to detect a difference in overall response rate of 28% at the end of 4 cycles of PAD. This is based on the assumptions that 44% of patients have amplification of 1q21 1, 2, the overall response rate with PAD combination therapy is 80%; the overall response rate with PAD if PAD therapy does not overcome 1q21 amplification is assumed to be 64%, while without 1q21 amplification it is assumed to be 92%. That is: Overall Response Rate (ORR) = P1q21 amplified x ORRamplified + P1q21 not amplified x ORRnot amplified i.e. 80% = 44% x 64% + 56% x 92%. The sample size of 105 allows for a 20% drop-out rate. Four 21-day cycles of PAD: a combination of bortezomib i.v. (intravenous) 1.3 mg/m2 (Days 1, 4, 8 and 11), doxorubicin i.v. 20 mg/m2 (days 1 and 4) and dexamethasone p.o. (by mouth) (days 1, 2, 4, 5, 8, 9, 11 and 12).

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with multiple myeloma
* eligible for autologous stem cell transplantation
* meets pre-treatment lab criteria (as defined within protocol).

Exclusion Criteria:

* Previously received treatment for multiple myeloma (including prior therapy with radiation or pulsed dexamethasone), except localised radiation to a solitary lesion or plasmacytomas or 4 days of corticosteroid therapy
* have a current diagnosis of smoldering multiple myeloma, monoclonal gammopathy of undetermined significance (MGUS), or Waldenström Macroglobulinemia
* have a history of any other malignancy within 5 years before enrolment
* have other significant comorbidities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-01; Primary Completion 2011-03 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Pty Ltd Clinical Trial, Study Director — Janssen-Cilag Pty Ltd
Locations (16):
- Australia (16):
  - Adelaide
  - Box Hill
  - Brisbane
  - Camperdown
  - Geelong
  - Gosford
  - Greenslopes
  - Malvern
  - Melbourne
  - Parkville
  - Perth
  - Sydney
  - Westmead
  - Woden
  - Wollongong
  - Woolloongabba

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were enrolled at multiple sites in Australia
Pre-assignment Details: 107 participants were enrolled and they all received the study treatment.
Groups:
- 1q21 Amplified: Participants with 1q21 amplification. Four 21-day cycles of bortezomib 1.3 mg/m2 intravenous (IV) on Days 1, 4, 8 and 11; plus doxorubicin 20 mg/m2 IV on Days 1 and 4; and dexamethasone 20 mg oral on Days 1, 2, 4, 5, 8, 9, 11 and 12.
- 1q21 Not Amplified: Participants without 1q21 amplification. Four 21-day cycles of bortezomib 1.3 mg/m2 intravenous (IV) on Days 1, 4, 8 and 11; plus doxorubicin 20 mg/m2 IV on Days 1 and 4; and dexamethasone 20 mg oral on Days 1, 2, 4, 5, 8, 9, 11 and 12.
- Failed/Missing Test: Participants who failed 1q21 test/had missing results for 1q21 test. Four 21-day cycles of bortezomib 1.3 mg/m2 intravenous (IV) on Days 1, 4, 8 and 11; plus doxorubicin 20 mg/m2 IV on Days 1 and 4; and dexamethasone 20 mg oral on Days 1, 2, 4, 5, 8, 9, 11 and 12.
Period: Completed PAD Induction
Arm/Group | 1q21 Amplified | 1q21 Not Amplified | Failed/Missing Test
Started | 26 (Received allocated treatment) | 72 (Received allocated treatment) | 9 (Received allocated treatment)
Completed | 21 (Completed PAD induction) | 68 (Completed PAD induction) | 9 (Completed PAD induction)
Not Completed | 5 | 4 | 0
Not completed — Patient choice | 0 | 1 | 0
Not completed — Disease progression | 0 | 2 | 0
Not completed — Adverse Event | 4 | 0 | 0
Not completed — Death | 1 | 1 | 0
Period: Primary Endpoint Analysis
Arm/Group | 1q21 Amplified | 1q21 Not Amplified | Failed/Missing Test
Started | 21 (Completed PAD induction) | 68 (Completed PAD induction) | 9 (Completed PAD induction)
Completed | 20 (participants analyzed) | 63 (participants analyzed) | 8 (participants analyzed)
Not Completed | 1 | 5 | 1
Not completed — Other | 1 | 2 | 0
Not completed — Patient choice | 0 | 1 | 0
Not completed — Efficacy data unavailable | 0 | 2 | 0
Not completed — Patient response missing | 0 | 0 | 1
Period: Completed 3-month Follow up
Arm/Group | 1q21 Amplified | 1q21 Not Amplified | Failed/Missing Test
Started | 20 (Participants analyzed for primary endpoint) | 63 (Participants analyzed for primary endpoint) | 8 (Participants analyzed for primary endpoint)
Completed | 20 (Completed 3-month follow-up) | 60 (Completed 3-month follow-up) | 8 (Completed 3-month follow-up)
Not Completed | 0 | 3 | 0
Not completed — Other | 0 | 2 | 0
Not completed — Physician Decision | 0 | 1 | 0
Period: Secondary Endpoint Analysis
Arm/Group | 1q21 Amplified | 1q21 Not Amplified | Failed/Missing Test
Started | 20 (Completed 3-month follow-up) | 60 (Completed 3-month follow-up) | 8 (Completed 3-month follow-up)
Completed | 20 (Participants analyzed for secondary endpoint) | 58 (Participants analyzed for secondary endpoint) | 7 (Participants analyzed for secondary endpoint)
Not Completed | 0 | 2 | 1
Not completed — Efficacy data unavailable | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1q21 Amplified | 1q21 Not Amplified | Failed/Missing Test | Total
Number analyzed (Participants) | 26 | 72 | 9 | 107
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (7.6) | 58.1 (10.1) | 55.6 (8.1) | 57.9 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 26 | 4 | 39
  Male | 17 | 46 | 5 | 68
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 23 | 63 | 8 | 94
  Asian | 1 | 2 | 0 | 3
  Mauritian | 1 | 0 | 0 | 1
  Indian | 0 | 1 | 0 | 1
  Middle Eastern | 0 | 0 | 1 | 1
  South American | 0 | 1 | 0 | 1
  Appears White | 1 | 4 | 0 | 5
  Missing race | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR): Number of Participants Who Are Responders (Had Stringent Complete Response [sCR], CR, Very Good Partial Response [VGPR] or Partial Response [PR]) After 4 Cycles of Bortezomib, Doxorubicin and Dexamethasone (PAD) Induction
Description: International Myeloma Working Group (IMWG) criteria - CR: negative immunofixation on the serum and urine, no soft tissue plasmacytomas and <5% plasma cells in the bone marrow; sCR: CR+normal free light chain ratio, no clonal cells in bone marrow by immunohistochemistry or immunofluorescence; VGPR: serum and urine M-protein detected by immunofixation but not electrophoresis, >90% in serum M-protein+urine, M-protein level <100 mg/24hour; PR: ≥50% decrease of serum and M-protein, 24 hour urinary M-protein decrease by ≥90% or <200 mg/24hour
Time Frame: 84 days
Population: Intent-to-treat (ITT) population- All enrolled participants who proceeded to receive Day 1 of Cycle 1 of PAD induction.
Measure: Number; unit: Participants
Groups:
- Total: Four 21-day cycles of bortezomib 1.3 mg/m2 intravenous (IV) on Days 1, 4, 8 and 11; plus doxorubicin 20 mg/m2 IV on Days 1 and 4; and dexamethasone 20 mg oral on Days 1, 2, 4, 5, 8, 9, 11 and 12.
Arm/Group | 1q21 Not Amplified | 1q21 Amplified | Failed/Missing Test | Total
Number analyzed (Participants) | 63 | 20 | 8 | 91
Participants
  Non Responder | 8 | 0 | 1 | 9
  Responder | 55 | 20 | 7 | 82
  Total | 63 | 20 | 8 | 91
Statistical Analysis 1: Comparison: 1q21 Not Amplified vs 1q21 Amplified; Null Hypothesis: There is no difference in response rate between 1q21 amplified and 1q21 NOT amplified; Test type: Superiority or Other; p = 0.09, Chi-squared

2. Secondary Outcome: Disease Response After 4 Cycles of Bortezomib, Doxorubicin and Dexamethasone (PAD) Induction
Description: Number of participants who achieved stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR) and stable disease (SD).
Time Frame: 84 days
Population: Intent-to-treat (ITT) population - All participants who were screened and received at least one dose of PAD
Measure: Number; unit: Particiipants
Groups:
- Failed/Missing: Participants who failed 1q21 test/had missing results for 1q21 test. Four 21-day cycles of bortezomib 1.3 mg/m2 intravenous (IV) on Days 1, 4, 8 and 11; plus doxorubicin 20 mg/m2 IV on Days 1 and 4; and dexamethasone 20 mg oral on Days 1, 2, 4, 5, 8, 9, 11 and 12.
Arm/Group | 1q21 Not Amplified | 1q21 Amplified | Failed/Missing | Total
Number analyzed (Participants) | 63 | 20 | 8 | 91
Particiipants
  stringent complete response (sCR) | 5 | 3 | 1 | 9
  complete response (CR) | 6 | 3 | 0 | 9
  Very Good Partial Response (VGPR) | 15 | 3 | 3 | 21
  Partial Response (PR) | 29 | 11 | 3 | 43
  Stable Disease (SD) | 8 | 0 | 1 | 9
  Total | 63 | 20 | 8 | 91
Statistical Analysis 1: Comparison: 1q21 Not Amplified vs 1q21 Amplified; Null Hypothesis: There is no difference in response rate between 1q21 amplified and 1q21 NOT amplified; Test type: Superiority or Other; p = 0.23, Chi-squared

3. Secondary Outcome: Overall Response Rate (ORR) to Bortezomib, Doxorubicin and Dexamethasone (PAD) Induction 3-months Following Autologous Stem Cell Transplant (ASCT).
Description: Responders are the number of participants who achieved stringent complete response (sCR)/ complete response (CR), very good partial response (VGPR) or partial response (PR) following PAD induction.
Time Frame: 3-months following ASCT
Population: Intent-to-treat (ITT) population - All participants who were screened and received at least one dose of PAD
Measure: Number; unit: Participants
Arm/Group | 1q21 Not Amplified | 1q21 Amplified | Failed/Missing | Total
Number analyzed (Participants) | 58 | 20 | 7 | 85
Participants
  Non Responder | 4 | 0 | 0 | 4
  Responder | 54 | 20 | 7 | 81
  Total | 58 | 20 | 7 | 85
Statistical Analysis 1: Comparison: 1q21 Not Amplified vs 1q21 Amplified; Null Hypothesis: There is no difference in response rate between 1q21 amplified and 1q21 NOT amplified; Test type: Superiority or Other; p = 0.23, Chi-squared

4. Secondary Outcome: Disease Response 3-months After Autologous Stem Cell Transplant (ASCT)
Description: Number of participants who achieved stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), stable disease (SD) and relapse as per IMWG criteria.
Time Frame: 3-months after ASCT
Population: Intent-to-treat (ITT) population - All participants who were screened and received at least one dose of PAD
Measure: Number; unit: Participants
Arm/Group | 1q21 Not Amplified | 1q21 Amplified | Failed/Missing | Total
Number analyzed (Participants) | 58 | 20 | 7 | 85
Participants
  stringent complete response (sCR) | 6 | 5 | 3 | 14
  complete response (CR) | 8 | 3 | 0 | 11
  Very Good Partial Response (VGPR) | 21 | 7 | 1 | 29
  Partial Response (PR) | 19 | 5 | 3 | 27
  Stable Disease (SD) | 3 | 0 | 0 | 3
  Relapse | 1 | 0 | 0 | 1
  Total | 58 | 20 | 7 | 85
Statistical Analysis 1: Comparison: 1q21 Not Amplified vs 1q21 Amplified; Null Hypothesis: There is no difference in response rate between 1q21 amplified and 1q21 NOT amplified; Test type: Superiority or Other; p = 0.56, Chi-squared

5. Secondary Outcome: Event Free Survival (EFS)
Description: Percentage of participants who did not have any of the following events: Death, Disease progression, Relapse, Cardiovascular accidents, Deep vein thrombosis, Pulmonary embolism, Fracture, Acute renal failure, Nervous system disorders 2 years after Day 1 Cycle 1 of bortezomib, doxorubicin and dexamethasone (PAD).
Time Frame: 2 years after Day 1 Cycle 1 of PAD
Population: Intent-to-treat (ITT) population - All participants who were screened and received at least one dose of PAD
Measure: Number; unit: Percentage of participants
Arm/Group | 1q21 Not Amplified | 1q21 Amplified
Number analyzed (Participants) | 58 | 20
Percentage of participants | 75.0 | 69.6
Statistical Analysis 1: Comparison: 1q21 Not Amplified vs 1q21 Amplified; Null Hypothesis: There is no difference in response rate between 1q21 amplified and 1q21 NOT amplified; Test type: Superiority or Other; p = 0.01, Log Rank

6. Secondary Outcome: Overall Survival
Description: Percentage of participants who had no event of death 2 years after Day 1 Cycle 1 of bortezomib, doxorubicin and dexamethasone (PAD).
Time Frame: 2 years after Day 1 Cycle 1 of PAD
Population: Intent-to-treat (ITT) population - All participants who were screened and received at least one dose of PAD
Measure: Number; unit: Percentage of participants
Arm/Group | 1q21 Not Amplified | 1q21 Amplified
Number analyzed (Participants) | 58 | 20
Percentage of participants | 93.8 | 86.4
Statistical Analysis 1: Comparison: 1q21 Not Amplified vs 1q21 Amplified; Null Hypothesis: There is no difference in response rate between 1q21 amplified and 1q21 NOT amplified; Test type: Superiority or Other; p = 0.28, Log Rank

7. Secondary Outcome: Assessment of Quality of Life (AQoL) Scores
Description: The AQoL is a multi-attribute utility health-related quality of life (HRQoL) instrument. It combines the 4 dimensions of independent living, relationships, senses and mental health into a single utility score. The AQoL instrument scores between 1 (best HRQoL) and -0.04 (worst possible HRQoL).
Time Frame: Up to 2 years
Population: Intent-to-treat (ITT) population - All participants who were screened and received at least one dose of PAD
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 1q21 Not Amplified | 1q21 Amplified | Failed/Missing | Total
Number analyzed (Participants) | 42 | 19 | 8 | 69
Scores on a scale | 0.0516596 (0.2769184) | 0.0068695 (0.3366162) | 0.1267145 (0.1839149) | 0.0480281 (0.2844673)

8. Secondary Outcome: Overall Response Rate (ORR) Stratified by Protein Expression (p53)
Description: Number of participants who are responders and nonresponders after 4 cycles of bortezomib, doxorubicin and dexamethasone (PAD) induction stratified by protein expression (p53).
Time Frame: 84 days
Population: Intent-to-treat (ITT) population - All participants who were screened and received at least one dose of PAD. The ORR was imputed, with those who discontinued treatment or who had efficacy data unavailable being coded as Non-Responders.
Measure: Number; unit: Participants
Groups:
- Negative: Participants without p53 expression
- Positive: Participants with p53 expression
Arm/Group | Negative | Positive
Number analyzed (Participants) | 75 | 14
Participants
  p53 Non Responder | 14 | 3
  p53 Responder | 61 | 11

9. Secondary Outcome: Overall Response Rate (ORR) Stratified by Protein Expression (Cyclin D1).
Description: Number of participants who are responders and nonresponders after 4 cycles of bortezomib, doxorubicin and dexamethasone (PAD) induction stratified by protein expression (Cyclin D1).
Time Frame: 84 days
Population: as for outcome 8
Measure: Number; unit: Participants
Groups:
- Negative: Participants without Cyclin D1 expression
- Positive: Participants with Cyclin D1 expression
Arm/Group | Negative | Positive
Number analyzed (Participants) | 59 | 25
Participants
  Cyclin D1 Non Responder | 11 | 5
  Cyclin D1 Responder | 48 | 20

10. Secondary Outcome: Overall Response Rate (ORR) Stratified by Protein Expression (Bcl-2)
Description: Number of participants who are responders and nonresponders after 4 cycles of bortezomib, doxorubicin and dexamethasone (PAD) induction stratified by protein expression (bcl-2)
Time Frame: 84 days
Population: as for outcome 8
Measure: Number; unit: Participants
Groups:
- Negative: Participants without bcl-2 expression
- Positive: Participants with bcl-2 expression
Arm/Group | Negative | Positive
Number analyzed (Participants) | 12 | 77
Participants
  bcl-2 Non Responder | 2 | 15
  bcl-2 Responder | 10 | 62

11. Secondary Outcome: Overall Response Rate (ORR) Stratified by Protein Expression (FGFR3)
Description: Number of participants who are responders and nonresponders after 4 cycles of bortezomib, doxorubicin and dexamethasone (PAD) induction stratified by protein expression (FGFR3)
Time Frame: 84 days
Population: as for outcome 8
Measure: Number; unit: Participants
Groups:
- Negative: Participants without FGFR3 expression
- Positive: Participants with FGFR3 expression
Arm/Group | Negative | Positive
Number analyzed (Participants) | 78 | 11
Participants
  FGFR3 Non Responder | 14 | 2
  FGFR3 Responder | 64 | 8

12. Secondary Outcome: Overall Survival (OS) Stratified by Protein Expression (p53).
Description: Percentage of participants who had no event of death 2 years after Day 1 Cycle 1 of bortezomib, doxorubicin and dexamethasone (PAD) stratified by protein expression (p53).
Time Frame: 2 years after Day 1 Cycle 1 of PAD
Population: Intent-to-treat (ITT) population - All participants who were screened and received at least one dose of PAD. The OS was not imputed.
Measure: Number; unit: Percentage of participants
Arm/Group | Negative | Positive
Number analyzed (Participants) | 65 | 13
Percentage of participants | 90.7 | 92.3

13. Secondary Outcome: Overall Survival (OS) Stratified by Protein Expression (Cyclin D1)
Description: Percentage of participants who had no event of death 2 years after Day 1 Cycle 1 of bortezomib, doxorubicin and dexamethasone (PAD) stratified by protein expression (Cyclin D1).
Time Frame: 2 years after Day 1 Cycle 1 of PAD
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | Negative | Positive
Number analyzed (Participants) | 49 | 24
Percentage of participants | 89.8 | 95.8

14. Secondary Outcome: Overall Survival (OS) Stratified by Protein Expression (Bcl-2)
Description: Percentage of participants who had no event of death 2 years after Day 1 Cycle 1 of bortezomib, doxorubicin and dexamethasone (PAD) stratified by protein expression (bcl-2).
Time Frame: 2 years after Day 1 Cycle 1 of PAD
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | Negative | Positive
Number analyzed (Participants) | 12 | 66
Percentage of participants | 91.7 | 90.9

15. Secondary Outcome: Overall Survival (OS) Stratified by Protein Expression (FGFR3)
Description: Percentage of participants who had no event of death 2 years after Day 1 Cycle 1 of bortezomib, doxorubicin and dexamethasone (PAD) stratified by protein expression (FGFR3).
Time Frame: 2 years after Day 1 Cycle 1 of PAD
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | Negative | Positive
Number analyzed (Participants) | 67 | 11
Percentage of participants | 92.5 | 81.8

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | 1q21 Amplified | 1q21 Not Amplified | Failed/Missing Test | Total
Serious Adverse Events (participants affected / at risk) | 15/26 | 30/72 | 5/9 | 50/107
Other Adverse Events (participants affected / at risk) | 26/26 | 72/72 | 9/9 | 107/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1q21 Amplified (N=26) | 1q21 Not Amplified (N=72) | Failed/Missing Test (N=9) | Total (N=107)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2
Atrial Fibrillation (Cardiac disorders) | 0 | 2 | 0 | 2
Cardiac Amyloidosis (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac Failure (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 1
Ventricular Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 6 | 0 | 6
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0 | 3
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 5 | 0 | 5
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Chest Pain (General disorders) | 0 | 2 | 0 | 2
Fatigue (General disorders) | 1 | 0 | 0 | 1
Gait Disturbance (General disorders) | 1 | 0 | 0 | 1
Oedema (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 5 | 2 | 9
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1
Device Related Infection (Infections and infestations) | 1 | 1 | 0 | 2
H1N1 Influenza (Infections and infestations) | 2 | 0 | 0 | 2
Herpes Zoster (Infections and infestations) | 0 | 1 | 1 | 2
Herpes Zoster Ophthalmic (Infections and infestations) | 0 | 1 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 5 | 0 | 5
Pneumonia (Infections and infestations) | 2 | 6 | 2 | 10
Pneumonia Viral (Infections and infestations) | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 2
Streptococcal Infection (Infections and infestations) | 0 | 1 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 2 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Urinary Retention Postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Blood Creatine Increased (Investigations) | 1 | 0 | 0 | 1
Blood Sodium Decreased (Investigations) | 0 | 1 | 0 | 1
Cardioactive Drug Level Increased (Investigations) | 0 | 1 | 0 | 1
Chest X-Ray Abnormal (Investigations) | 0 | 1 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 5 | 0 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 6
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Autonomic Neuropathy (Nervous system disorders) | 0 | 2 | 0 | 2
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 2
Facial Palsy (Nervous system disorders) | 0 | 1 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 1 | 2 | 0 | 3
Presyncope (Nervous system disorders) | 0 | 2 | 0 | 2
Syncope (Nervous system disorders) | 1 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Acute Febrile Neutrophilic Dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pain Management (Surgical and medical procedures) | 1 | 0 | 0 | 1
Circulatory Collapse (Vascular disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 1 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1q21 Amplified (N=26) | 1q21 Not Amplified (N=72) | Failed/Missing Test (N=9) | Total (N=107)
Anaemia (Blood and lymphatic system disorders) | 8 | 15 | 3 | 26
Neutropenia (Blood and lymphatic system disorders) | 6 | 12 | 0 | 18
Vision Blurred (Eye disorders) | 2 | 6 | 2 | 10
Abdominal Pain (Gastrointestinal disorders) | 2 | 5 | 1 | 8
Constipation (Gastrointestinal disorders) | 17 | 42 | 6 | 65
Diarrhoea (Gastrointestinal disorders) | 9 | 26 | 3 | 38
Dyspepsia (Gastrointestinal disorders) | 3 | 9 | 1 | 13
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4 | 7 | 0 | 11
Nausea (Gastrointestinal disorders) | 10 | 36 | 5 | 51
Reflux Gastritis (Gastrointestinal disorders) | 1 | 5 | 0 | 6
Vomiting (Gastrointestinal disorders) | 1 | 15 | 1 | 17
Chest Pain (General disorders) | 1 | 8 | 0 | 9
Fatigue (General disorders) | 7 | 30 | 4 | 41
Mucosal Inflammation (General disorders) | 2 | 7 | 1 | 10
Oedema (General disorders) | 3 | 4 | 0 | 7
Oedema Peripheral (General disorders) | 5 | 12 | 2 | 19
Pain (General disorders) | 1 | 8 | 1 | 10
Pyrexia (General disorders) | 1 | 5 | 1 | 7
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 9 | 0 | 11
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 8 | 1 | 9
Decreased Appetite (Metabolism and nutrition disorders) | 4 | 11 | 1 | 16
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 4 | 0 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 3 | 0 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 4 | 0 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 15 | 0 | 18
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1 | 6
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 | 5 | 0 | 9
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 9 | 0 | 10
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 8 | 1 | 14
Areflexia (Nervous system disorders) | 2 | 6 | 1 | 9
Dizziness (Nervous system disorders) | 1 | 14 | 1 | 16
Dysgeusia (Nervous system disorders) | 8 | 14 | 3 | 25
Headache (Nervous system disorders) | 4 | 14 | 0 | 18
Lethargy (Nervous system disorders) | 6 | 11 | 0 | 17
Neuralgia (Nervous system disorders) | 3 | 14 | 1 | 18
Neuropathy Peripheral (Nervous system disorders) | 15 | 36 | 3 | 54
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 16 | 1 | 18
Anxiety (Psychiatric disorders) | 3 | 5 | 0 | 8
Insomnia (Psychiatric disorders) | 9 | 27 | 3 | 39
Mood Altered (Psychiatric disorders) | 2 | 5 | 1 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 11 | 4 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 10 | 0 | 16
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 2 | 9
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 20 | 2 | 25
Rash (Skin and subcutaneous tissue disorders) | 8 | 11 | 1 | 20
Orthostatic Hypotension (Vascular disorders) | 3 | 6 | 0 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days